CLINICAL TRIAL: NCT02830672
Title: Comparative Clinical Study of Ultrasound-Guided A1 Pulley Release vs Open Surgical Intervention in the Treatment of Trigger Finger
Brief Title: Ultrasound Guided A1 Pulley Release For The Treatment of Trigger Finger
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Vasileios S. Nikolaou, Assistant Professor Of Orthopedics, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Surgical Release of Ai Pulley Trigger Finger

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open surgical release A1 Pulley (Active Comparator)
  Interventions: Procedure: Surgical release A1 pulley for Trigger finger of the hand
- Ultrasound guided close release A1 pulley (Active Comparator)
  Interventions: Procedure: Surgical release A1 pulley for Trigger finger of the hand

INTERVENTIONS:
Procedure: Surgical release A1 pulley for Trigger finger of the hand

SUMMARY:
In this randomized, prospective clinical trial, patients with trigger finger or trigger thumb, will be treated with two different methods; ultrasound-guided release of the first annular pulley or open surgical release of A1 pulley. Results will be compared regarding functional, clinical and cosmetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resistant -after conservative treatment- trigger finger or trigger thumb, suffering at least for 3 months.

Exclusion Criteria:

* Patients under 18 years old, these who were treated with a previous operation or a corticosteroid injection for their disease and those who were suffering by inflammatory arthritis, tumor or autoimmune disease.
* Patients with multiple trigger fingers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Resolution of triggering expressed as the "success rate" per digit. | 12 weeks

SECONDARY OUTCOMES:
The time for taking postoperative pain killers | 12 weeks
Range of motion recovery | 12 weeks
QuickDASH test scores (Greek version) | 12 weeks
Time to return to normal activities (including work) | 12 weeks
Cosmetic results | 12 weeks

IPD SHARING:
Plan to Share IPD: No